CLINICAL TRIAL: NCT02757339
Title: Evaluating the Neurobiological Basis of Traumatic Dissociation in a Cross-Diagnostic Sample of Women With Histories of Childhood Abuse and Neglect
Brief Title: Evaluating the Neurobiological Basis of Traumatic Dissociation in Women With Histories of Abuse and Neglect
Status: Enrolling by invitation | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Milissa Kaufman, Director of The Dissociative Disorders and Trauma Research Program, Mclean Hospital
Other Study IDs: 2014P001429
Record Dates: First submitted 2016-03-17; First posted 2016-05-02 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorders; Dissociative Identity Disorder
Keywords: neurobiology; PTSD; DID
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Dissociative Identity Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Study participants will provide a 2mm saliva sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with History of Childhood Abuse: The study will enroll up to 140 female patients with either DID or PTSD ages 18-89
- Healthy Control Group: We will recruit up to 60 control subjects matched for demographics (age, race, gender).

SUMMARY:
This study aims to evaluate the neurobiological basis of traumatic dissociation in a cross-diagnostic sample of women who have histories of childhood abuse and neglect.

DETAILED DESCRIPTION:
Dissociative symptoms commonly are associated with exposure to traumatic stress. Preliminary evidence from functional magnetic resonance imaging-based analysis (fMRI) of neural activation during dissociative symptom provocation in patients with PTSD or DID has implicated certain key structures involved in the generation of dissociative symptoms. Given the presumed region-to-region neural interplay implicit within this model, the investigators believe the use of intrinsic functional connectivity MRI (fcMRI) represents a valuable next line of investigation into the neurobiology of traumatic dissociation. The investigators also believe that a genetic approach holds promise as another converging line of inquiry into our understanding of traumatic dissociation.

To evaluate the neurobiological basis of traumatic dissociation, this study will recruit patients with PTSD or DID, and recruit matched controls to identify neurobiological correlates of traumatic dissociation.The study will compare the phenomenology of traumatic dissociation in patients with different PTSD subtypes and DID using standardized measures to look at the neurological and genetic correlates.

This study will also include a follow up visit that includes neuroimaging and genetic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Clinical diagnosis of PTSD or DID and history of childhood abuse, or healthy controls
* Age between 18 and 89
* Legal and mental competency of the patient

Exclusion Criteria:

* Male
* Under 18 or over 89
* Legal or mental incompetence
* Delirium secondary to medical illness
* PTSD or DID due to general medical or neurological illness
* History of neurological conditions that may cause significant psychiatric symptomatology (e.g., dementia)
* Any contraindication to MR scans, including claustrophobia, pregnancy, metal implants, etc.
* Current alcohol or substance dependence or abuse (within the last month)
* A history of schizophrenia or other psychotic disorder
* History of head injury or loss of consciousness for longer than 5 min (including concussion)

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 90 female patients with either DID or PTSD ages 18-89. We will also recruit up to 60 control subjects matched for demographics (age, race, gender).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline correlates of traumatic dissociation in Functional Magnetic Resonance Imaging at 36 to 56 weeks | Baseline and 36 to 56 weeks after baseline
  Study participation will involve a baseline 60 minute cognitive assessment and a 60 minute Magnetic Resonance Imaging (MRI) at the 3 Tesla magnet in the McLean Hospital Imaging Center focusing on attention, emotion regulation, and symptoms of depersonalization. The first time point is baseline.The second time point will be 36-56 weeks after the baseline 60 minute Magnetic Resonance Imaging (MRI) scan at the 3 Tesla magnet in the McLean Hospital Imaging Center.

CONTACTS AND LOCATIONS:
Overall Officials: Milissa L Kaufman, M.D./Ph.D, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided